CLINICAL TRIAL: NCT00894855
Title: Skin Cancer Screening and Education Program at Beaches
Brief Title: Skin Cancer Screening and Education at Beaches
Acronym: SHADE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: The Shilling SHADE Foundation of America (Unknown); University of Massachusetts, Amherst (Other); Harvard Medical School (HMS and HSDM) (Other); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Karen Emmons, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 14598
Record Dates: First submitted 2009-05-06; First posted 2009-05-07 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Skin Cancer
Keywords: skin cancer prevention; SHADE; Beach
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- education only (Active Comparator): This comprehensive education program included a health educator visit, on the education van, who gave education about sun safety.
  Interventions: Behavioral: education about sun protection
- education plus dermatologist skin exam (Experimental): In addition to the education program, participants received free skin exams by board certified dermatologists from Brigham and Women's Hospital. The van was equipped with a private clinical setting conducive to carry out such examinations. Based on the recommendations of the American Academy of Dermatology (AAD), a visual full body exam was provided to participants. At the end of each skin exam the dermatologist provided a presumptive diagnosis to the participant, and made appropriate recommendations and referrals for follow up with the participants' physician/dermatologist (if and when necessary). All participants undergoing the skin exam were required to complete an "AAD Skin Cancer Screening Registration and Report form".
  Interventions: Other: dermatologist skin exam
- educ, biometric fb, and derm skin exam (Experimental): Participants received the active components of the other three conditions.
  Interventions: Behavioral: biometric feedback; Other: dermatologist skin exam
- education plus biometric feedback (Experimental): In addition to the educational program, participants received biometric feedback using a Dermascan Analyzer and Ultra Violet (UV) Reflectance Photography. The Dermascan Analyzer is an educational tool that enhances visibility of skin texture, markings or lesions and is commonly used in health fairs and at schools all over the country. The analyzer highlights the sun damage on the participants skin as dark purple blotches, which the participants are able to see in the mirror placed inside the analyzer. Ultra Violet (UV) Reflectance Photography provides participants with a visual image of their skin damage that can be taken with them.
  Interventions: Behavioral: biometric feedback

INTERVENTIONS:
Behavioral: education about sun protection — This comprehensive education program included a visit with a health educator, on the education van, who gave education about sun safety.
  Arms: education only
Behavioral: biometric feedback — Participants received biometric feedback using a Dermascan Analyzer and Ultra Violet (UV) Reflectance Photography. The Dermascan Analyzer is an educational tool that enhances visibility of skin texture, markings or lesions and is commonly used in health fairs and at schools all over the country. The analyzer highlights the sun damage on the participants skin as dark purple blotches, which the participants are able to see in the mirror placed inside the analyzer. Ultra Violet (UV) Reflectance Photography provides participants with a visual image of their skin damage that can be taken with them.
  Arms: educ, biometric fb, and derm skin exam; education plus biometric feedback
Other: dermatologist skin exam — Full body skin exam.
  Arms: educ, biometric fb, and derm skin exam; education plus dermatologist skin exam

SUMMARY:
This study was an evaluation of the Dana-Farber Cancer Institute Blum Family Resource Center Van's existing skin cancer screening and education program. This program occurred over 2 summers. This study will fill a critical gap in the investigators' knowledge about how best to address the high-risk behaviors that regularly occur during the summertime at beaches. The investigators randomized beaches to receive different combinations of the van program components in order to determine how services should optimally be configured to maximize impact. The investigators hypothesized that providing all three components (1-Skin cancer prevention education; 2-Biometric feedback using a Dermascan Analyzer that illustrates skin damage due to sun exposure and Ultra Violet (UV) Reflectance Photography; and 3-Dermatologist skin exam) will maximize knowledge and behavior change, relative to education alone.

ELIGIBILITY:
Inclusion Criteria:

* Beachgoers eligible to participate in the study included:

  * those who were 18 years and older
  * Caucasian
  * able to understand, speak and read English
  * ability to give informed consent
  * had not already enrolled in the study at another participating beach

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 634 (Actual)
Dates: Start 2007-01; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
sun protection behaviors | 4-6 months post-intervention
sun burns | 4-6 months post-intervention
skin self-exams | 4-6 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Karen M Emmons, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States